CLINICAL TRIAL: NCT00028769
Title: Phase II Evaluation of Early Oral Estramustine, Oral Etoposide and Intravenous Paclitaxel in Combination With Hormone Therapy in Patients With High-Risk Metastatic Adenocarinoma of the Prostate
Brief Title: S0032, Combination Chemotherapy Plus Hormone Therapy in Treating Patients With Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069132; S0032 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2002-01-04; First posted 2003-01-27 (Estimated); Results first posted 2013-07-16 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-06

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Estramustine; Etoposide; Flutamide; Goserelin; Leuprolide; nilutamide; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hormone therapy, estramustine, etoposide and paclitaxel (Experimental): Hormone therapy (leuprolide, bicalutamide, nilutamide, goserelin, flutamide), estramustine, etoposide and paclitaxel
  Interventions: Drug: bicalutamide; Drug: estramustine; Drug: etoposide; Drug: flutamide; Drug: goserelin; Drug: leuprolide; Drug: nilutamide; Drug: paclitaxel

INTERVENTIONS:
Drug: bicalutamide
Drug: estramustine
  Other Names: estramustine phosphate sodium
Drug: etoposide
Drug: flutamide
Drug: goserelin
Drug: leuprolide
  Other Names: leuprolide acetate
Drug: nilutamide
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Androgens can stimulate the growth of prostate cancer cells. Drugs such as goserelin, leuprolide, flutamide, or bicalutamide may stop the adrenal glands from producing androgens. Combining chemotherapy with hormone therapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy plus hormone therapy in treating patients who have metastatic prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the progression-free and overall survival in patients with high-risk metastatic adenocarcinoma of the prostate treated with early estramustine, etoposide, and paclitaxel with combined androgen-blockade therapy.
* Determine the type, frequency, and severity of toxicity of this regimen in this patient population.

OUTLINE: This is a multicenter study.

* Androgen-blockade therapy: Patients receive a standard regimen of luteinizing hormone-releasing hormone agonist therapy comprising either goserelin subcutaneously once monthly or once every 3 months or leuprolide intramuscularly once monthly, once every 3 months, or once every 4 months. Patients also receive a standard regimen of antiandrogen therapy comprising oral bicalutamide, oral flutamide, or oral nilutamide once daily. Treatment continues in the absence of disease progression or unacceptable toxicity.
* Chemotherapy: Beginning 14-30 days after initiation of androgen-blockade therapy, patients receive oral estramustine three times daily and oral etoposide once daily on days 1-14 and paclitaxel IV over 1 hour on day 2. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months until disease progression, every 6 months for 2 years, and then annually for 3 years.

PROJECTED ACCRUAL: A total of 80 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed high-risk adenocarcinoma of the prostate

  * Clinical stage D2 disease as evidenced by one of the following:

    * Visceral disease (liver, lung, or other viscera)
    * Bone metastases to sites in both the axial (spine, pelvis, ribs, or skull) and appendicular (claviculae, humeri, or femora) skeleton
* No prior or concurrent (treated or untreated) brain metastases

  * Patients with clinical evidence of brain metastasis must have a negative brain CT or MRI
* No evidence of untreated spinal cord compression

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* Zubrod 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* No active hypercoagulability

Hepatic:

* Not specified

Renal:

* Not specified

Cardiovascular:

* No transient ischemic attacks, stroke, or myocardial infarction within the past 6 months
* No active coronary artery disease requiring antianginal therapy
* No active thrombophlebitis

Pulmonary:

* No history of pulmonary embolus

Other:

* No other prior malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or adequately treated stage I or II cancer currently in complete remission

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior biologic therapy and recovered
* No concurrent biologic therapy

Chemotherapy:

* No prior cytotoxic chemotherapy
* No other concurrent chemotherapy

Endocrine therapy:

* Prior androgen-blockade therapy (e.g., luteinizing hormone-releasing hormone agonist and antiandrogen therapy) allowed if administered for a duration of less than 30 days
* Prior neoadjuvant hormonal therapy allowed

Radiotherapy:

* At least 4 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy

Surgery:

* At least 4 weeks since prior surgery and recovered

Other:

* No concurrent bisphosphonates

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2001-12; Primary Completion 2010-06 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C. Smith, MD, Study Chair — University of Michigan Rogel Cancer Center
Locations (91):
- United States (91):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Carl T. Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock, Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Veterans Affairs Medical Center - West Los Angeles, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - University of California Davis Cancer Center, Sacramento, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - MBCCOP - Howard University Cancer Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Tampa (Haley), Tampa, Florida
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago Westside Hospital, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines, Hines, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane Cancer Center at Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Health System, Detroit, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - Saint Louis University Cancer Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Western New York Urology Associates, Cheektowaga, New York
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Veterans Affairs Medical Center - Charleston, Charleston, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - University of Tennessee Cancer Institute at Methodist Central Hospital, Memphis, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Texas Tech University Health Sciences Center School of Medicine, Amarillo, Texas
  - Veterans Affairs Medical Center - Amarillo, Amarillo, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - UMC Southwest Cancer and Research Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - Sentara Cancer Institute at Sentara Norfolk General Hospital, Norfolk, Virginia
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - Puget Sound Oncology Consortium, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- CAD + Chemo: Patients receive Combined androgen deprivation (CAD) therapy with LHRH agonist (goserelin acetate or leuprolide acetate) sq/IM q 1-4 months depending on dose chosen by the treating physician and oral antiandrogen (250 mg/tid of flutamide, 50 mg/d of bicalutamide or 300 mg/d for 30 days then 150 mg/d of nilutamide) given continuously until disease progression and Chemotherapy (4 cycles of estramustine 280 mg orally 3 times daily and etoposide 50 mg/m^2 daily for 14 days of each 21-day cycle, with paclitaxel 135 mg/m^2 given intravenously within 1 hour on day 2 of each cycle)
Period: Overall Study
Arm/Group | CAD + Chemo
Started | 41
Eligible | 36
Eligible and Began Protocol Therapy | 35 (One patient refused all protocol treatment and was not evaluable for the present analysis)
Completed | 0 (Patients receive protocol treatments until evidence of disease progression)
Not Completed | 41
Not completed — Adverse Event | 2
Not completed — Refusal Unrelated to Adverse Events | 1
Not completed — Progression or Death | 31
Not completed — Other - Not Protocol Specified | 1
Not completed — Ineligible | 5
Not completed — Not Analyzable | 1

BASELINE CHARACTERISTICS:
Arm/Group | CAD + Chemo
Number analyzed (Participants) | 35
Age Continuous [Median (Full Range); unit: years] | 60 [45 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Southwestern Oncology Group Performance Status [Number; unit: participants] — Patients will be graded according to the Zubrod performance status scale. 0: Fully active, able to carry all pre-disease performance without restriction. 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature. 2: Ambulatory and capable of self-care but unable to carry out any work activities; up and about more than 50% of waking hours. 3: Capable of limited self-care, confined to bed or chair more than 50% of waking hours. 4: Completely disabled; cannot carry on any self-care; totally confined to bed or chair.
  participants
    0 | 20
    1 | 15
Bone Pain Grade (CTC version 2.0) [Number; unit: participants] — 0 - none, 1 - mild pain not interfering with function, 2 - moderate pain: pain or analgesics interfering with function, but not interfering with activities of daily living, 3 - severe pain: pain or analgesics severely interfering with activities of daily living, 4 - disabling
  participants
    Missing | 2
    <2 | 26
    >=2 | 7
Previous Prostatectomy [Number; unit: participants]
  Yes | 6
  No/Unknown | 29
Gleason Score [Number; unit: participants]
  Missing | 1
  6 | 2
  7 | 12
  8 | 6
  9-10 | 14

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Measured from time of registration to time of first documentation of progression determined from the prostate-specific antigen (PSA) level, clinical criteria, or symptomatic deterioration. PSA progression is defined as a 25% increase greater than baseline. If the patient's PSA level had decrease during the study, a 25% increase from the nadir PSA level, with absolute value of >=5 ng/mL is considered progression. CLinical progress is defined as the appearance of any new lesion at any site or death without documented progression. Symptomatic deterioration is defined as a global deterioration of the health status requiring discontinuation of treatment without objective evidence of progression.
Time Frame: 0-5 years (assessed every 3 months if no progression when the chemotherapy had been finished. Once off chemotherapy, assessed every 3 months until progression)
Population: All eligible patients who started treatment were included in the analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CAD + Chemo
Number analyzed (Participants) | 35
months | 13 [10 to 16]

2. Secondary Outcome: Number of Patients With Grade 3 Through Grade 5 Adverse Events That Are Related to Study Drug
Description: Adverse Events (AEs) are reported by the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 2.0. For each patient, worst grade of each event type is reported. Grade 3 = Severe, Grade 4 = Life-threatening, Grade 5 = Fatal.
Time Frame: up to 5 years after registration
Population: Eligible patients who had received any treatment were included in the adverse event summaries. Any CTCAE 2.0 event of Grade 3 (severe), Grade 4 (life threatening), or Grade 5 (fatal) which deemed to be related to protocol treatment are included.
Measure: Number; unit: Participants
Arm/Group | CAD + Chemo
Number analyzed (Participants) | 35
Participants
  Alkaline phosphatase increase | 1
  Anemia | 1
  Bilirubin increase | 1
  Cardiac ischemia/infarction | 1
  Confusion | 1
  Constipation/bowel obstruction | 1
  Edema | 2
  Erectile impotence | 3
  Fatigue/malaise/lethargy | 2
  GI-other | 1
  Hyperglycemia | 2
  Infection w/o 3-4 neutropenia | 1
  Infection with 3-4 neutropenia | 2
  Leukopenia | 9
  Lymphopenia | 2
  Neutropenia/granulocytopenia | 9
  PRBC transfusion | 2
  Pain-other | 1
  Prothrombin time increase | 1
  Renal failure | 1
  Second primary | 1
  Thrombocytopenia | 1
  Thrombosis/embolism | 4

3. Primary Outcome: Overall Survival (OS)
Description: Overall survival is defined from the date of registration to date of death from any cause
Time Frame: 0-5 years
Population: All eligible patients who started treatment were included in the analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CAD + Chemo
Number analyzed (Participants) | 35
months | 38 [28 to 49]

ADVERSE EVENTS:
Time Frame: Patients were assessed for adverse events after every cycle (1 cycle = 21 days) of protocol treatment
Arm/Group | CAD + Chemo
Serious Adverse Events (participants affected / at risk) | 6/35
Other Adverse Events (participants affected / at risk) | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CAD + Chemo (N=35)
Cardiac ischemia/infarction (Cardiac disorders) | 2
Flu-like symptoms-other (General disorders) | 1
Infection with 3-4 neutropenia (Infections and infestations) | 1
Abnormal troponin I (cTnI) (Investigations) | 1
Leukopenia (Investigations) | 1
Second primary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thrombosis/embolism (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CAD + Chemo (N=35)
Anemia (Blood and lymphatic system disorders) | 18
PRBC transfusion (Blood and lymphatic system disorders) | 2
Abdominal pain/cramping (Gastrointestinal disorders) | 2
Constipation/bowel obstruction (Gastrointestinal disorders) | 6
Diarrhea without colostomy (Gastrointestinal disorders) | 8
Dyspepsia/heartburn (Gastrointestinal disorders) | 3
Esophagitis/dysphagia (Gastrointestinal disorders) | 3
GI-other (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 20
Proctitis (Gastrointestinal disorders) | 4
Stomatitis/pharyngitis (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 9
Edema (General disorders) | 12
Fatigue/malaise/lethargy (General disorders) | 30
Fever without neutropenia (General disorders) | 3
Pain-other (General disorders) | 15
Infection w/o 3-4 neutropenia (Infections and infestations) | 3
Respiratory infect w/o neutrop (Infections and infestations) | 3
Alkaline phosphatase increase (Investigations) | 5
Bilirubin increase (Investigations) | 4
Creatinine increase (Investigations) | 2
Leukopenia (Investigations) | 21
Lymphopenia (Investigations) | 4
Neutropenia/granulocytopenia (Investigations) | 13
SGOT (AST) increase (Investigations) | 11
SGPT (ALT) increase (Investigations) | 3
Thrombocytopenia (Investigations) | 3
Weight gain (Investigations) | 4
Weight loss (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 6
Hyperglycemia (Metabolism and nutrition disorders) | 10
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 6
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 4
Joint,muscle,bone-other (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Myalgia/arthralgia, NOS (Musculoskeletal and connective tissue disorders) | 2
Dizziness/light headedness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 5
Sensory neuropathy (Nervous system disorders) | 8
Weakness (motor neuropathy) (Nervous system disorders) | 4
Confusion (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 8
Dysuria (Renal and urinary disorders) | 3
Hematuria (Renal and urinary disorders) | 5
Incontinence (Renal and urinary disorders) | 3
Urinary frequency/urgency (Renal and urinary disorders) | 5
Urinary retention (Renal and urinary disorders) | 3
Erectile impotence (Reproductive system and breast disorders) | 8
Gynecomastia (Reproductive system and breast disorders) | 6
Libido loss (Reproductive system and breast disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 18
Nail changes (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash/desquamation (Skin and subcutaneous tissue disorders) | 5
Skin-other (Skin and subcutaneous tissue disorders) | 3
Hot flashes (Vascular disorders) | 9
Hypertension (Vascular disorders) | 2
Thrombosis/embolism (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No